CLINICAL TRIAL: NCT00521001
Title: A Phase II Study of Temozolomide and Everolimus (RAD001) Therapy for Metastatic Melanoma
Brief Title: Temozolomide and Everolimus in Treating Patients With Stage IV Melanoma That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0675; NCI-2012-02713 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000562166 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Everolimus; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- everolimus + temozolomide (Experimental): Patients receive oral everolimus once a day on days 1-5, 8-12, 15-19, 22-26, and 29-33 and oral temozolomide once a day on days 8-12 for course 1 only. For course 2 and all subsequent courses, patients receive oral everolimus once a day on days 1-5, 8-12, 15-19, and 22-26 and oral temozolomide once a day on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  All patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for relative numbers of T, B, and NK cells via flow cytometry, quantitative immunoglobulin levels (IgG, IgM, and IgA), Tetramer/ELISPOT CTL frequencies to CMV/EBV immunodominant antigens, V beta T cell spectratyping, and VEGF levels via ELISA.
  After completion of study treatment, patients are followed every 8 weeks.
  Interventions: Drug: everolimus; Drug: temozolomide

INTERVENTIONS:
Drug: everolimus
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. Giving everolimus together with temozolomide may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving everolimus together with temozolomide works in treating patients with stage IV melanoma that cannot be removed by surgery

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the 9-week progression-free survival rate for patients with stage IV malignant melanoma treated with everolimus and temozolomide.

Secondary

* Evaluate overall survival time.
* Evaluate time to disease progression.
* Evaluate confirmed response rate.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once a day on days 1-5, 8-12, 15-19, 22-26, and 29-33 and oral temozolomide once a day on days 8-12 for course 1 only. For course 2 and all subsequent courses, patients receive oral everolimus once a day on days 1-5, 8-12, 15-19, and 22-26 and oral temozolomide once a day on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

All patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for relative numbers of T, B, and NK cells via flow cytometry, quantitative immunoglobulin levels (IgG, IgM, and IgA), Tetramer/ELISPOT CTL frequencies to CMV/EBV immunodominant antigens, V beta T cell spectratyping, and VEGF levels via ELISA.

After completion of study treatment, patients are followed every 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma with manifestations of metastatic disease.
* Unresectable stage IV malignant melanoma with measurable disease

  * Measurable disease defined as at least one lesion with the longest diameter measured as ≥ 20 mm by CT scan or MRI scan OR ≥ 10 mm by spiral CT
* No previously untreated or unstable active brain metastases within the past 3 months
* No known standard therapy for this disease that is potentially curative or proven capable of extending life expectancy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9.0 g/dL
* Alkaline phosphatase ≤ 3 times institutional upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* AST ≤ 3 times ULN
* INR ≤ 1.5
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients and their partners must use effective contraception during and for ≥ 8 weeks after completion of study treatment
* Able to return to a NCCTG institution for follow-up
* Able to forego foods high in fat content 2 hours prior to and 2 hours after administration of everolimus therapy
* Able to provide blood samples for research purposes
* No hypersensitivity to temozolomide, dacarbazine, or any analog of sirolimus
* No history of malignancy within the past 5 years except for basal cell or squamous cell carcinoma of the skin treated with local resection only
* No immunosuppression from any cause, including known HIV infection or chronic immunosuppressive therapy
* No impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome)
* No serious medical condition that may make it unsafe for a patient to enroll in study, including any of the following:

  * Severely impaired lung function (FEV1 < 1 liter), unstable angina pectoris (ongoing symptoms), ongoing symptomatic congestive heart failure (i.e., NYHA class I-IV) refractory to appropriate therapy, or myocardial infarction within the past 6 months, or serious uncontrolled cardiac arrhythmia
  * Uncontrolled diabetes in spite of optimal therapy (i.e., a history of fasting serum glucose > 150 mg/dL)
  * Any active (acute or chronic) or uncontrolled infection/disorders
  * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the study treatment
  * Liver disease (i.e., uncompensated cirrhosis or active hepatitis with elevated liver enzymes)
* No bleeding diathesis
* No concurrent severe condition that would make it undesirable for the patient to participate in this trial or that would jeopardize compliance with the trial

PRIOR CONCURRENT THERAPY:

* Must have recovered from effects of prior antineoplastic therapy
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas)
* At least 4 weeks since prior immunotherapy
* At least 4 weeks since prior biologic therapy
* At least 4 weeks since prior radiosurgery
* At least 4 weeks since prior investigational therapy for melanoma
* No prior small bowel resection that may significantly alter the absorption of everolimus
* No prior sirolimus or its analogues
* No prior radiotherapy to > 30% of bone marrow
* No concurrent drugs that may induce CYP3A4 activity
* No concurrent warfarin
* No concurrent grapefruit or grapefruit juice
* No concurrent use or planned use of vaccines containing live virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi D. Rao, MD, MBBS, Study Chair — Mayo Clinic
Locations (198):
- United States (198):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Dronca RS, Allred JB, Perez DG, Nevala WK, Lieser EA, Thompson M, Maples WJ, Creagan ET, Pockaj BA, Kaur JS, Moore TD, Marchello BT, Markovic SN. Phase II study of temozolomide (TMZ) and everolimus (RAD001) therapy for metastatic melanoma: a North Central Cancer Treatment Group study, N0675. Am J Clin Oncol. 2014 Aug;37(4):369-76. doi: 10.1097/COC.0b013e31827b45d4. PMID 23357973

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus + Temozolomide: Patients receive 10 mg everolimus orally once a day on days 1-5, 8-12, 15-19, 22-26, and 29-33 and 200 mg/m^2 temozolomide orally once a day on days 8-12 for cycle 1 only (where cycle length is 35 days). For cycle 2 and all subsequent cycles, patients receive 10 mg everolimus orally once a day on days 1-5, 8-12, 15-19, and 22-26 and 200 mg/m^2 temozolomide orally once a day on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Everolimus + Temozolomide
Started | 49
Completed | 48
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus + Temozolomide
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 60 [29 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: 9-week Progression-free Survival Rate
Description: The primary endpoint of this trial is the 9 week PFS rate. A patient is a success if they are progression free at their cycle 2 evaluation (approximately 9 weeks post registration). All patients, who meet the eligibility criteria, sign a consent form, and start treatment will be included in the evaluation of the 9-week PFS rate (evaluable patients). The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated using the properties of the binomial distribution. If some patients are lost to follow up prior to their cycle 2 evaluation, the Kaplan-Meier method will be used to estimate the 9 week PFS rate. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: at 9 weeks
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Everolimus + Temozolomide
Number analyzed (Participants) | 48
proportion of patients | 0.44 [0.29 to 0.59]

2. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause; Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Temozolomide
Number analyzed (Participants) | 48
months | 8.6 [7.1 to 12.2]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to the earliest date documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. The distribution of time to progression will be estimated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from registration to the earliest date documentation of disease progression; Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Temozolomide
Number analyzed (Participants) | 48
months | 2.4 [2.1 to 4.0]

4. Secondary Outcome: Confirmed Response Rate (Complete Response and Partial Response)
Description: Confirmed response rates will be evaluated by dividing the number of confirmed responders (i.e. patients that achieve a CR or PR on consecutive evaluations) by the total number of evaluable patients. Confidence intervals for the true response rate will be calculated using the properties of the binomial distribution.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of confirmed responses
Arm/Group | Everolimus + Temozolomide
Number analyzed (Participants) | 48
percentage of confirmed responses | 8.3 [2.3 to 20.0]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed within 14 days prior to registration and during the Active Monitoring Phase at the start of each treatment cycle; Up to 5 years.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for AE reporting. All graded adverse events are reported.
Arm/Group | Everolimus + Temozolomide
Serious Adverse Events (participants affected / at risk) | 6/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus + Temozolomide (N=48)
Palpitations (Cardiac disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 4 (4)
Platelet count decreased (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus + Temozolomide (N=48)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (14)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 19 (27)
Nausea (Gastrointestinal disorders) | 27 (40)
Vomiting (Gastrointestinal disorders) | 13 (16)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 39 (116)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 31 (90)
Lymphocyte count decreased (Investigations) | 27 (101)
Neutrophil count decreased (Investigations) | 22 (43)
Platelet count decreased (Investigations) | 21 (58)
Serum cholesterol increased (Investigations) | 4 (8)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 21 (39)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (6)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (22)
Taste alteration (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (20)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes